CLINICAL TRIAL: NCT02361216
Title: Efficacy and Safety of Ingenol Mebutate Gel in Field Treatment of Actinic Keratosis on Full Face, Balding Scalp or Approximately 250 cm2 on the Chest
Brief Title: Efficacy and Safety of Ingenol Mebutate Gel for Actinic Keratosis Applied on Large Area on Face, Scalp or Chest
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LP0105-1032
Record Dates: First submitted 2015-02-02; First posted 2015-02-11 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2018-10

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingenol mebutate gel (Experimental): Treatment once daily for 3 days
  Interventions: Drug: Ingenol Mebutate
- Vehicle (Placebo Comparator): Treatment once daily for 3 days
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: Ingenol Mebutate
  Arms: Ingenol mebutate gel
Other: Vehicle — Vehicle gel
  Arms: Vehicle

SUMMARY:
The objective of the trial is to investigate efficacy and safety of ingenol mebutate gel for actinic keratosis applied to large treatment areas once daily for three consecutive days on face, scalp or chest.

ELIGIBILITY:
Inclusion Criteria:

Subjects with 5 to 20 clinically typical, visible and discrete, actinic keratosis (AKs) non-hyperkeratotic and non-hypertrophic AKs within a selected treatment area of sun-damaged skin on either:

* The full face
* The full balding scalp
* A contiguous area of approximately 250 cm2 on the chest

Exclusion Criteria:

* Location of the treatment area (full face, full balding scalp or chest) within 5 cm of an incompletely healed wound or within 5 cm of a suspected basal cell carcinoma (BCC) or squamous cell carcinoma (SCC).
* Previously assigned treatment in this clinical trial or previously participated in a clinical trial in the LEO clinical programme on ingenol mebutate gel for larger treatment areas.
* Treatment with ingenol mebutate gel in the selected treatment area within the last 12 months.
* Lesions in the treatment area that have: atypical clinical appearance (e.g. cutaneous horn) and/or, recalcitrant disease (e.g., did not respond to cryotherapy on two previous occasions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. William Hanke, MD, Principal Investigator — Laser & Skin Surgery Center of Indiana,
Locations (1):
- Laser & Skin Surgery Center of Indiana, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were followed for 8 weeks following the first application of investigational medicinal product (IMP) at Day 1 (3-day treatment period including an 8-week follow-up period) and for an additional 12 months following Week 8 (extended 12-month follow-up period).
Groups:
- Ingenol Mebutate Gel: Treatment once daily for 3 days
  Ingenol mebutate gel 0.027% or vehicle gel was applied on either the full face, full balding scalp, or within a contiguous area of approximately 250 cm2 on the chest.
- Vehicle Gel: Treatment once daily for 3 days
  Vehicle: Vehicle gel
Period: 3 Day Treatment and 8 Week Follow/up
Arm/Group | Ingenol Mebutate Gel | Vehicle Gel
Started | 552 | 177
Completed | 541 | 158
Not Completed | 11 | 19
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Unacceptable Local Skin Reaction (LSR) | 1 | 0
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Trial site closed | 3 | 3
Not completed — Lost to Follow-up | 0 | 2
Period: 12-month Follow-up
Arm/Group | Ingenol Mebutate Gel | Vehicle Gel
Started | 541 | 157 (1 of the 158 subjects did not receive treatment and was also excluded from the 12-month follow-up.)
Completed | 489 | 130
Not Completed | 52 | 27

BASELINE CHARACTERISTICS:
Groups:
- Ingenol Mebutate Gel: Treatment once daily for 3 days
  Ingenol Mebutate
- Total: Total of all reporting groups
Arm/Group | Ingenol Mebutate Gel | Vehicle | Total
Number analyzed (Participants) | 552 | 177 | 729
Age, Continuous [Median (Full Range); unit: years] | 68 [38 to 91] | 69 [45 to 91] | 68 [38 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 45 | 194
  Male | 403 | 132 | 535
Region of Enrollment [Number; unit: participants]
  United States | 304 | 98 | 402
  Canada | 188 | 59 | 247
  Australia | 60 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Actinic Keratosis (AK)
Description: Complete resolution of actinic keratosis (AKclear100) at Week 8 is defined as 100% reduction from baseline in the number of clinically visible AKs
Time Frame: 8 weeks
Population: Of the 729 subjects randomised to treatment, 4 did not receive treatment. These 4 subjects (3 subjects in active treatment group and 1 in vehicle group) were excluded from the Full Analysis Set (FAS), which consisted of 725 subjects (549 subjects in active treatment group and 176 in corresponding vehicle group). AKclear100 is based on the FAS
Measure: Number; unit: percentage of participants
Groups:
- Ingenol Mebutate Gel: Treatment once daily for 3 days with ingenol mebutate with 8 week follow-up after initial treatment
- Vehicle: Treatment once daily for 3 days vehicle gel with 8 week follow-up after initial treatment
Arm/Group | Ingenol Mebutate Gel | Vehicle
Number analyzed (Participants) | 549 | 176
percentage of participants | 21.4 | 3.4
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel vs Vehicle; AKclear100 at Week 8: full analysis set. The null hypothesis was that there is no difference at Week 8 in AKclear100 rates between ingenol mebutate gel 0.027% and vehicle gel. This hypothesis was tested against the 2-sided alternative of a difference between the 2 treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Ratio of clearance rates = 6.29, 95% CI 2-sided [2.82 to 14]

2. Secondary Outcome: Percentage of Participants With Partial Clearance at Week 8
Description: Partial clearance (AKclear75 ) is defined as a reduction in the number of clinically visible AKs in the selected treatment area by at least 75% compared to baseline.
Time Frame: 8 weeks
Population: AKclear75 at Week 8 is based on the full analysis set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol Mebutate Gel | Vehicle
Number analyzed (Participants) | 549 | 176
percentage of participants | 59.4 | 8.9
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel vs Vehicle; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The prespecified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Ratio of clearance rates = 6.81, 95% CI 2-sided [4.16 to 11.1] — Mantel-Haenszel estimate (0.027% relative to vehicle), adjusted for pooled sites

3. Secondary Outcome: Percentage of Participants With Partial Clearance at Week 4
Description: Partial clearance (AKclear75) defined as a reduction in the number of clinically visible AKs in the selected treatment area by at least 75% compared to baseline.
Time Frame: 4 weeks
Population: AKclear75 at Week 4 is based on the full analysis set (FAS)
Measure: Number; unit: percentage of participants
Arm/Group | Ingenol Mebutate Gel | Vehicle
Number analyzed (Participants) | 549 | 176
percentage of participants | 59.8 | 9.2
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel vs Vehicle; The p-values for secondary endpoints have been corrected by the Holm-Bonferroni method to account for multiplicity. The pre-specified multiplicity adjustment by the Holm-Bonferroni method requires the ordering of the p-values for the secondary endpoints by size; Test type: Superiority or Other; p < 0.001, Mantel Haenszel; Ratio of clearance rates = 6.53, 95% CI 2-sided [4.04 to 10.5]

4. Secondary Outcome: Percent Reduction From Baseline in AK Count
Description: Percent reduction in AK count in the selected treatment area at Week 8
Time Frame: 8 weeks
Population: Percent reduction in AK count is based on the full analysis set (FAS)
Measure: Mean (95% Confidence Interval); unit: percentage reduction of AK count
Groups:
- Vehicle Gel: Treatment once daily for 3 days vehicle gel with 8 week follow-up after initial treatment
Arm/Group | Ingenol Mebutate Gel | Vehicle Gel
Number analyzed (Participants) | 549 | 176
percentage reduction of AK count | 75.7 [73.9 to 77.3] | 12.7 [3.0 to 21.4]
Statistical Analysis 1: Comparison: Ingenol Mebutate Gel vs Vehicle Gel; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Negative binominal regression with log baseline count as offset variable and treatment group, anatomical location stratum and pooled site as factors; Ratio of clearance = 0.28, 95% CI 2-sided [0.24 to 0.32]

ADVERSE EVENTS:
Time Frame: 14 Months
Description: A total of 729 subjects were randomised to treatment, of whom 4 did not receive treatment with IMP. These 4 subjects (3 subjects from the active treatment group and 1 from the corresponding vehicle group) were excluded from the Full Analysis Set, which consisted of 725 subjects (549 subjects in the active treatment group and 176 in the corresponding vehicle group).
  The Safety Analysis Set was the same as the Full Analysis Set.
Arm/Group | Ingenol Mebutate Gel | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/549 | 0/176
Serious Adverse Events (participants affected / at risk) | 8/549 | 2/176
Other Adverse Events (participants affected / at risk) | 394/549 | 18/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel (N=549) | Vehicle (N=176)
Myocardial Infarction (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ingenol Mebutate Gel (N=549) | Vehicle (N=176)
Application Site Pain (General disorders) | 350 | 4
Application Site Pruritus (General disorders) | 203 | 7
Application Site Discomfort (General disorders) | 28 | 2
application site parasthesia (General disorders) | 14 | 2
headache (Nervous system disorders) | 22 | 4
eyelid oedema (Eye disorders) | 14 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes